CLINICAL TRIAL: NCT02443974
Title: Effectiveness of Knee Bracing in Elderly With Knee Osteoarthritis: a Randomized, Controlled Trial
Brief Title: Bracing to Treat Knee Osteoarthritis in Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Christine Brumini, MsC, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP 1248/09
Record Dates: First submitted 2015-04-08; First posted 2015-05-14 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Braces

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Knee brace group (Experimental): Patients received knee brace with hinges (Fisiotensor®) and were instructed to use it in daily activities, every day, during six months
  Interventions: Device: Brace (Fisiotensor®)
- Knee sleeve group (Experimental): Patients received knee sleeve without hinges (Fisiotensor®) and were instructed to use it in daily activities, every day, during six months
  Interventions: Device: Sleeve (Fisiotensor®)
- Control group (No Intervention): Keep medication usual

INTERVENTIONS:
Device: Brace (Fisiotensor®)
  Arms: Knee brace group
Device: Sleeve (Fisiotensor®)
  Arms: Knee sleeve group

SUMMARY:
Background: Osteoarthritis (OA) is highly prevalent in the elderly, with the knee being the most commonly affected joint in this population. Knee braces are often used to prevent common problems in knees during daily activities. The purpose of these devices is to decrease pain and improve functionality. In the literature some studies have tested the effectiveness of unloader brace for valgus or varus. However, the braces most used in the investigators' clinical setting and the less costly ones have not been described in quality studies in the literature. There are only few studies on this subject and they are methodologically inadequate. There are no studies that compared the effectiveness between the knee brace with metal hinges (no alignment) and knee brace without metal hinges. Objective: To evaluate the effectiveness of knee braces on pain, function and quality of life in the elderly with knee OA. Methods: Elderly with knee OA, both genders, with pain scale 3-7cm on a 10cm pain numeric scale were included. Of the 222 patients screened, 120 met the eligibility criteria and were randomized to the groups: without metal hinges, with metal hinges or control group. The groups without and with metal hinges received knee brace and were instructed to use it in daily activities, every day, during three months. Assessment for pain (NPS), function (WOMAC and Knee Lequesne) and quality of life (SF-36) were done at baseline and after 45, 90 and 180 days by a blinded assessor.

ELIGIBILITY:
Inclusion Criteria:

* pain in numerical pain scale between 3 and 7cm;
* Knee ligamentous instability

Exclusion Criteria:

* fibromyalgia and neurologic disease;
* knee or hip replacement
* surgery scheduled in the following 6 months
* start physical activity or received joint injection in the past three months
* need to use walking aids or brace in knee

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in pain measured by a numeric pain scale | Baseline, after 45, 90 and 180 days

SECONDARY OUTCOMES:
Change in function measured by Lequesne and WOMAC questionnaires | Baseline, after 45, 90 and 180 days
Change in quality of life measured by SF-36 questionnaire | Baseline, after 45, 90 and 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No